CLINICAL TRIAL: NCT07348224
Title: Pharmacokinetics and Pharmacodynamics of Synthetic Nicotine and Nicotine Analogues
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Swiss Tobacco Prevention Funds (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: BASEC-ID 2025-01893
Record Dates: First submitted 2025-11-24; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Nicotine; Vaping; Synthetic Nicotine; Nicotine Analogues
Keywords: synthetic nicotine; nicotine analogues; vaping
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Synthetic S-Nicotine (Other): Vaping of e-liquids contanining synthetic S-nicotine
  Interventions: Other: Vaping of synthetic S-nicotine
- Racemic nicotine (S-/R-nicotine) (Other): Vaping of e-liquids contanining synthetic racemic nicotine (containing both the S- and R-nicotine enantiomers)
  Interventions: Other: Vaping of racemic nicotine (S-/R-nicotine)
- 6-methylnicotine (Other): Vaping of e-liquids contanining the nicotine analogue 6-methylnicotine (6MN)
  Interventions: Other: Vaping of 6-methylnicotine

INTERVENTIONS:
Other: Vaping of synthetic S-nicotine — Vaping of e-liquids containing synthetic S-nicotine
  Arms: Synthetic S-Nicotine
Other: Vaping of racemic nicotine (S-/R-nicotine) — Vaping of e-liquids containing synthetic racemic nicotine (S-/R-nicotine)
  Arms: Racemic nicotine (S-/R-nicotine)
Other: Vaping of 6-methylnicotine — Vaping of e-liquids containing the nicotine analogue 6-methylnicotine (6MN)
  Arms: 6-methylnicotine

SUMMARY:
Electronic cigarettes are battery-operated devices that can produce an aerosol by heating a liquid which commonly contains nicotine. In recent years, products containing synthetically produced nicotine and nicotine analogues have entered the market. However, it remains unclear whether these types of nicotine have the same effects as conventional nicotine derived from the tobacco plant. The aim of this study is to investigate the effects of these nicotine types and to gain a better understanding of their respective mechanisms of action.

DETAILED DESCRIPTION:
In the first part of the study, participants will use electronic cigarettes containing synthetic nicotine or nicotine analogs at three sessions in the hospital, following a specific schedule. In the second part, each product will be used for four days outside the hospital. The study is double-blind, meaning neither the participants nor the study team will know which product is being used.

The study comprises a total of seven appointments at the hospital. During these appointments, participants will be asked questions about their electronic cigarette and tobacco use, and samples of saliva, urine, and blood will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, age 18 or older at screening who have used EC with nicotine during at least 10 of the past 30 days
* Saliva cotinine concentration of > 30 ng/mL at screening
* Ability to communicate well with the investigator and to understand and comply with the requirements of the study
* Women of child-bearing age engaging in sexual activities which can lead to pregnancy: willingness of using a reliable/hormonal contraception method during the study (hormonal, e.g. pill, intrauterine devices, or mechanical method, e.g. condom, diaphragm)
* Signed informed consent form

Exclusion Criteria:

* Known hypersensitivity/allergy to a content of the e-liquids
* Smoking of more than 5 cigarettes per day in the past 30 days
* Pregnant or lactating women
* Intention to become pregnant during the course of the study
* BMI < 18 or > 30 kg/m2 at screening
* History or clinical evidence of alcoholism or drug abuse within the 3-year period prior to screening
* Loss of ≥ 250 mL of blood within 3 months prior to screening, including blood donation
* Treatment with an investigational drug within 30 days prior to screening
* Treatment with prescribed or over-the-counter medications with known influence on CYP2A6 function within 1 week prior to screening (with the exception of contraception)
* History or clinical evidence of any disease (e.g. gastrointestinal tract-disease) and/or existence of any surgical or medical condition, which in the opinion of the investigator might interfere with the absorption, distribution, metabolism or excretion of the study drugs, or which might increase the risk of toxicity.
* Legal incapacity or limited legal capacity at screening
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum total nicotine concentrations (Cmax) | 15 minutes before vaping and 2, 5, 15, 30, 60, 120, and 180 minutes after the last puff
  Comparison of the maximum total nicotine (i.e. sum of both enantiomers) in blood concentrations (Cmax) between groups

SECONDARY OUTCOMES:
Maximum concentration (Cmax) of 6-methylnicotine | 15 minutes before vaping and 2, 5, 15, 30, 60, 120, and 180 minutes after the last puff
  Maximum concentration of 6-methylnicotine in blood
Maximum concentration (Cmax) of 6-methylnicotine's metabolites | 15 minutes before vaping and 2, 5, 15, 30, 60, 120, and 180 minutes after the last puff
  Maximum concentration of 6-methylnicotine's metabolites in blood
AUC (area under the concentration-time curve) nicotine enantiomers | 15 minutes before vaping and 2, 5, 15, 30, 60, 120, and 180 minutes after the last puff
  Area under the concentration-time curve (AUC) of nicotine enantiomers in blood
AUC (area under the concentration-time curve) 6-methylnicotine | 15 minutes before vaping and 2, 5, 15, 30, 60, 120, and 180 minutes after the last puff
  Area under the concentration-time curve (AUC) of 6-methylnicotine in blood
AUC (area under the concentration-time curve) 6-methylnicotine's metabolites | 15 minutes before vaping and 2, 5, 15, 30, 60, 120, and 180 minutes after the last puff
  Area under the concentration-time curve (AUC) of 6-methylnicotine's metabolites in blood
Tmax (time of Cmax) nicotine enantiomers | 15 minutes before vaping and 2, 5, 15, 30, 60, 120, and 180 minutes after the last puff
  Tmax of nicotine enantiomers in blood
Tmax (time of Cmax) 6-methylnicotine | 15 minutes before vaping and 2, 5, 15, 30, 60, 120, and 180 minutes after the last puff
  Tmax of 6-methylnicotine in blood
Tmax (time of Cmax) 6-methylnicotine's metabolites | 15 minutes before vaping and 2, 5, 15, 30, 60, 120, and 180 minutes after the last puff
  Tmax of 6-methylnicotine's metabolites in blood
T1/2 (elimination half-life) nicotine enantiomers | 15 minutes before vaping and 2, 5, 15, 30, 60, 120, and 180 minutes after the last puff
  Elimination half-life (T1/2) of nicotine enantiomers in blood
T1/2 (elimination half-life) 6-methylnicotine | 15 minutes before vaping and 2, 5, 15, 30, 60, 120, and 180 minutes after the last puff
  Elimination half-life (T1/2) of 6-methylnicotine in blood
T1/2 (elimination half-life) 6-methylnicotine's metabolites | 15 minutes before vaping and 2, 5, 15, 30, 60, 120, and 180 minutes after the last puff
  Elimination half-life (T1/2) of 6-methylnicotine's metabolites in blood
Blood nicotine metabolite ratio (NMR) | 15 minutes before vaping
  Nicotine clearance assessed using the 3'-hydroxycotinine/cotinine ratio (i.e. nicotine metabolite ratio (NMR)
Saliva nicotine metabolite ratio (NMR) | At baseline
  Nicotine clearance assessed using the 3'-hydroxycotinine/cotinine ratio (i.e. nicotine metabolite ratio (NMR)
Blood steroid hormone levels | At baseline, 15 minutes before vaping and 2, 5, 15, 30, 60, 120, and 180 minutes after the last puff during the first part of the study and following 4 days ad libitum use during the second part
  Steroid hormone levels in blood
Saliva steroid hormone levels | At baseline
  Steroid hormone levels in saliva
Urine steroid hormone levels | At baseline and following 4 days ad libitum use of each product
  Steroid hormone levels in urine
Heart rate | Baseline, 15 minutes before vaping and 2, 5, 15, 30, 60, 120, and 180 minutes after the last puff, at study completion (2.5-6.5 weeks after screening)
  bpm
Blood pressure | Baseline, 15 minutes before vaping and 2, 5, 15, 30, 60, 120, and 180 minutes after the last puff, at study completion (2.5-6.5 weeks after screening)
  mmHg
Modified Minnesota Nicotine Withdrawal Scale (MNWS) | Baseline, 10 minutes, 1 hour and 3 hours after last puff
  Score/questionnaire asssessing withdrawal: The Modified Minnesota Nicotine Withdrawal Scale (MNWS) (excluding items related to sleep disturbance and constipation) including eight items (angry/irritable/frustrated, anxious/nervous, depressed mood/sad, desire or craving to smoke, difficulty concentrating, increased appetite/hungry, restless and impatient), rated on a 0=none to 4=severe scale.
Tiffany Questionnaire on Smoking Urges-Brief (QSU) total (global) craving score | Baseline, 10 minutes, 1 hour and 3 hours after last puff
  Score/questionnaire asssessing craving: The Tiffany Questionnaire on Smoking Urges-Brief (QSU) total (global) craving score as the average of all responses (mean of ten items, rated on a 1=strongly disagree to 7=strongly agree scale).
Positive and Negative Affect Schedule (PANAS) | Baseline, 10 minutes, 1 hour and 3 hours after last puff
  Score/questionnaire asssessing satisfaction: The Positive and Negative Affect Schedule (PANAS) including items assigned as Positive or Negative Affect (each score is the sum of ten items, rated on a 1=very slightly/not at all to 5=extremely scale).
Respiratory symptoms | Baseline and 5 minutes after last puff
  Questions regarding shortness of breath, wheezing, cough, phlegm; posisble answers: yes/no
Direct effects | 10 minutes post-use
  Questions regarding e.g. satisfying, calming, pleasant, vape another one right now, using visual analog scales (0-100 mm) with a single word scored from left (not at all) to right (extremely).
Modified e-cigarette evaluation questionnaire (mCEQ) | Following 4 days ad libitum use of each product
  Questionnaire asssessing subjective effects
Urinary total nicotine equivalents (TNE) concentrations | Following 4 days ad libitum use of each product
  Molar sum of urinary total (parent and glucuronide) nicotine, cotinine and 3'-hydroxycotinine
Urinary volatile organic compounds (VOC) concentrations | Following 4 days ad libitum use of each product
  VOC in urine

OTHER OUTCOMES:
Reported adverse events | Throughout study completion, an average of 2.5-6.5 weeks
  Classification and severity grading scale in accordance with the "Common Terminology Criteria for Adverse Events CTCAE Version 5.0" terminology.

CONTACTS AND LOCATIONS:
Locations (1):
- Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided